CLINICAL TRIAL: NCT05899673
Title: A Phase 3, Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Fazirsiran in Participants With Alpha-1 Antitrypsin Deficiency-Associated Liver Disease
Brief Title: An Extension Study to Learn About the Long-Term Safety of Fazirsiran and if Fazirsiran Can Help People With Alpha-1 Antitrypsin Liver Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-999-3003; 2023-503497-21-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Alpha1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fazirsiran 200 mg (Experimental): Participants who are currently taking part in or who have completed their treatment in parent studies AROAAT2001 (NCT03945292) and AROAAT2002 (NCT03946449) may rollover in this study to receive fazirsiran, 200 milligrams (mg), injection, subcutaneously on Day 1 and once every 12 weeks (Q12W) thereafter until fazirsiran receives approval and is commercially available in the participant's country, until a participant withdraws from the study or the sponsor decides to terminate the study.
  Interventions: Drug: Fazirsiran Injection

INTERVENTIONS:
Drug: Fazirsiran Injection — Fazirsiran will be injected subcutaneously.
  Other Names: TAK-999; ARO-AAT

SUMMARY:
The main aim of this study is to learn if fazirsiran is safe during long-term use in people with liver disease caused by the abnormal Z-alpha-1 antitrypsin (Z-AAT) protein. People who have taken part in previous fazirsiran studies (AROAAT2001 [NCT03945292] or AROAAT2002 [NCT03946449]) can continue to receive fazirsiran every 3 months as long as they participate in this study, the study is ongoing or until health authorities in their country approve fazirsiran to be publicly available. The study may also provide information on whether fazirsiran has a long-term effect in reducing liver fibrosis or slowing down the progression of liver fibrosis in people with liver disease due to the abnormal Z-AAT protein.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be eligible for inclusion in the study:
* The participant is willing and able to understand and fully comply with study procedures and requirements, in the opinion of the investigator.
* The participant is able to read, understand, and complete the study questionnaires electronically per investigator's judgment.
* The participant has provided informed consent (ICF) (that is, in writing, documented via a signed and dated ICF) and any required privacy authorization before the initiation of any study procedures.

Note: For participants who comprehend, can provide informed consent, and are unable to sign the ICF, an impartial witness may sign the ICF on behalf of the participant after the participant has orally consented to the participant's participation in the study.

* The participant enrolling in this open-label extension (OLE) study will have participated in a previously qualifying study, and will be considered for eligibility based on the following study-specific criteria:
* AROAAT2001:

  * Participants with fibrosis may roll over into this OLE study after they reach their next regularly scheduled, Q12W visit.
  * Participants with fibrosis who have completed the AROAAT2001 study may be enrolled into the OLE study.
* AROAAT2002:

  * Participants in Cohorts 1 and 1b may roll over after completing the 24-week primary study period.
  * Participants in Cohort 2 may roll over after completing the 48-week primary study period.
  * Participants who have completed the study may be enrolled into the OLE study.
* The participant is a nonsmoker (defined as: does not smoke cigarettes daily for at least 24 weeks) with current nonsmoking status confirmed by urine cotinine at Day 1.

  * E-cigarettes (vapor) are not permitted.
  * The participant may be on nicotine replacement (patch or gum). A positive urine cotinine result due to nicotine replacement is acceptable for enrollment at the discretion of the investigator.
* The participant must have suitable venous access for blood sampling.
* It must be confirmed that the participant does not have hepatocellular carcinoma (HCC). Participants will be screened for HCC with alpha-fetoprotein (AFP) and abdominal ultrasound. If the participant has any of the following, they will be required to have contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) imaging to exclude HCC before enrollment.

  * AFP >20 nanogram per milliliter (ng/mL).
  * AFP 15 to 19 ng/mL at enrollment if that is >2 times prestudy levels (if available).
  * Any liver lesion >10 millimeter (mm) (longest diameter) detected by ultrasound.
  * Poor visibility of liver on ultrasound.
* A person of childbearing potential (POCBP) must have a negative urine pregnancy test performed within 3 days prior to Day 1 dosing in this study (sensitive to 25 International Unit [IU] human chorionic gonadotropin [hCG]).
* The participant must use appropriate contraception methods (that is, highly effective methods for female and medically appropriate methods for male study participants) for the entire duration of the study. Participants who terminate early must use appropriate contraception methods for 6 months after the last dose of study intervention. Male participants who terminate early must not donate sperm for at least 6 months after the last dose of study intervention.
* Sexual abstinence, for the purposes of this study, is only considered a highly effective method of contraception when considered to align with the preferred and usual lifestyle of the participant. It will be employed for the entire duration of the study and the 6 months after last dose of study intervention.
* Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea methods are not considered "true" abstinence and are not acceptable methods of contraception.

Exclusion Criteria:

* The participant will be excluded from the study if any of the following exclusion criteria are met:
* The participant is likely to require major surgery. Major surgery typically requires at least 1 night in the hospital. Examples include laparoscopic surgery (except cholecystectomy and tubal ligation); Gastrointestinal tract (GI) tract surgery including 1 or more segments of the colon or terminal ileum; open resection of organs; large joint replacements; mastectomy with reconstruction; and spine, thoracic, vascular, or intracranial surgery.
* The participant has evidence of other forms of chronic liver diseases, including viral hepatitis B or C, primary biliary cholangitis, primary sclerosing cholangitis, Wilson disease, alcoholic hepatitis, hemochromatosis, liver cancer, history of biliary diversion, or autoimmune hepatitis.
* The participant has abnormal finding(s) of clinical relevance during the evaluation before the first study dosing that, in the opinion of the investigator, could adversely impact participant safety during the study or adversely impact study results. For US only: Participants with baseline emphysema may be allowed into the OLE if their lung disease has been stable.
* The participant had major protocol deviation(s) in AROAAT2001 or AROAAT2002 that would affect the conduct of this study.
* The participant permanently discontinued investigational product because of an AE, adjudicated as related to the study intervention, in AROAAT2001 or AROAAT2002.
* Female participants who became pregnant during Study AROAAT2001 or AROAAT2002, female participants who are lactating or planning to become pregnant during the study period; or males or female participants of childbearing potential not agreeing to continue using appropriate contraception methods through the conclusion of study participation.
* The participant has a Child-Turcotte-Pugh (CTP) score >=7 OR (Model for End-Stage Liver Disease) MELD score >14.
* The participant meets Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Creatinine criteria as per the protocol. All laboratory tests used as exclusion criteria may be repeated once and the repeat value may be used for study eligibility determination.
* Participants who have a newly-diagnosed malignancy or recurrence of malignancy (except for resected cutaneous basal cell carcinoma, squamous cell carcinoma, superficial bladder tumors, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence).
* The participant is experiencing a pulmonary exacerbation at the time of enrollment (participant enrollment may be temporarily delayed after the clinical resolution of an exacerbation).
* The participant has unstable, poorly controlled, or severe hypertension. Participants may be reevaluated once their blood pressure is successfully controlled.
* The participant has a history of more than moderate alcohol consumption within 12 months before the Day 1 visit.
* The participant has a history of hypersensitivity or allergies to fazirsiran or any associated excipients.
* The participant has any concomitant medical or psychiatric condition or social situation that would make it difficult to comply with protocol requirements or put the participant at additional safety risk.
* The participant has a history of clinically significant hematologic, renal, hepatic, cardiovascular, infectious, pulmonary, neurologic, psychiatric, GI, systemic inflammatory, metabolic, or endocrine disorder or any other condition that, in the opinion of the investigator, rendered the participant a poor candidate for inclusion into the study.
* The participant has a history of thromboembolic disease (including deep vein thrombosis or pulmonary embolism), within 24 weeks before enrollment; or is taking chronic anticoagulants. (Note: Participants taking stable doses of chronic anticoagulants may be allowed after consultation with the medical monitor, if they do not have cirrhosis or a history of liver decompensating events).
* The participant is unable to return for all scheduled study visits.
* The participant has known or suspected coronavirus disease 2019 (COVID-19) that in the opinion of the sponsor and investigator does not resolve during screening. Positive antibody testing for COVID-19 without other evidence of current or recent active infection does not exclude participation. Enrollment of participants who fail inclusion due to COVID-19 infection may be temporarily delayed at the discretion of the sponsor and investigator. If the participant has a positive polymerase chain reaction (PCR) with no other evidence of infection, a retest may be allowed; however, to enroll in the study the participant must have a negative PCR.
* The participant is a study site employee, an immediate family member (for example, spouse, parent, child, sibling), or is in a dependent relationship with a study site employee who is involved in conduct of this study, or may consent under duress.
* The participant who, in the opinion of the investigator or the sponsor, will be uncooperative or unable to comply with study procedures.
* The participant who participates in other studies involving an investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2033-05-02 (Estimated); Study Completion 2033-05-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | From start of study drug administration (in current study) up to End of study (EOS) (current study [up to 10 years])
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not it is considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study intervention. An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, suspected transmission of any infectious agent, an important medical event. AEs and SAEs including any pulmonary AEs or SAEs indicative of worsening pulmonary condition (example, pulmonary exacerbation, respiratory infection, significant pulmonary function test decline) will be reported.
Number of Participants With Clinically Significant Changes From Baseline in Pulmonary Function Parameters | Baseline (current study), up to EOS (current study up to 10 years])
  Standard pulmonary function parameters measured will be used to study lung function. Clinical significance of pulmonary function parameters will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in Vital Signs | From start of study drug administration (in current study) up to EOS (current study [up to 10 years])
  Vital signs include body temperature, respiratory rate, sitting blood pressure (systolic and diastolic, resting more than 5 minutes), pulse, oxygen saturation. Clinical significance of vital signs will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in Laboratory Parameters | From start of study drug administration (in current study) up to EOS (current study [up to 10 years])
  Laboratory parameters include hematology, biochemistry including liver tests, coagulation, and urinalysis. Clinical significance of laboratory parameters will be determined at the investigator's discretion.

SECONDARY OUTCOMES:
Number of Participants With no Progression from Baseline of At least 1 Stage of Histologic Fibrosis on Liver Biopsy at Week 102 | At Week 102 (current study)
  Number of participants with no progression from baseline of at least 1 stage of histologic fibrosis (by Meta-Analysis of Histological Data in Viral Hepatitis [METAVIR] staging) on liver biopsy at Week 102 will be reported.
Number of Participants With Reduction from Baseline of At least 1 Stage of Histologic Fibrosis on Liver Biopsy at Week 102 | At Week 102 (current study)
  Number of participants with baseline fibrosis of F1 or higher, a decrease from baseline of at least 1 stage of histologic fibrosis (by METAVIR staging) on liver biopsy at Week 102 will be reported.
Change from Baseline in Intrahepatic Z-AAT Protein Polymer Burden Assessed by Periodic Acid Schiff Plus Diastase (PAS+D) Staining in Liver Biopsy at Week 102 | Baseline (current study), Week 102 (current study)
  Change from baseline in intrahepatic Z-AAT protein polymer burden assessed by PAS+D staining in liver biopsy will be assessed.
Change from Baseline in Intrahepatic Portal Inflammation Score at Week 102 in Liver Biopsy | Baseline (current study), Week 102 (current study)
  Change in portal inflammation score in liver biopsy, based on pathology slide reads. Inflammation will be assessed on a scale of 0-3, with higher scores showing more severe inflammation.
Change from Baseline in Liver Stiffness Assessed by Magnetic Resonance Elastography (MRE) | Baseline (current study), up to EOS (current study up to 10 years])
  Change from baseline in MRE-derived liver stiffness will be assessed.
Change from Baseline in Liver Stiffness Assessed by Vibration-Controlled Transient Elastography (VCTE) | Baseline (current study), up to EOS (current study up to 10 years])
  Change from baseline in VCTE-derived liver stiffness will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (5):
  - UCSD Altman Clinical and Translational Research Institute, La Jolla, California
  - Stanford Medicine Outpatient Center, Redwood City, California
  - UF Clinical and Translational Science Institute, Gainesville, Florida
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Medical University of South Carolina - Hollings Cancer Center - PPDS, Charleston, South Carolina
- Medizinische Universitat Wien (Medical University of Vienna), Vienna, Austria
- Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia, Germany
- Hospital Nélio Mendonça, Funchal, Portugal
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - Royal Infirmary of Edinburgh - PPDS, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/9e52333653b14cfe?idFilter=%5B%22TAK-999-3003%22%5D